CLINICAL TRIAL: NCT05497869
Title: Effects of Active Release Technique (ART) on Pectoralis Minor Tightness in Post Mastectomy Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Shafaq
Record Dates: First submitted 2022-08-10; First posted 2022-08-11 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Postgastrectomy Syndrome
Keywords: Pectoralis minor tightness; post mastectomy women; active release technique; breast cancer
MeSH Terms: conditions — Postgastrectomy Syndromes; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental interventional group (Experimental): Active Release Technique (ART)
  Interventions: Other: active release group
- active control group (Active Comparator): conventional group
  Interventions: Other: active control group

INTERVENTIONS:
Other: active release group — Patient is in supine lying position with 15-20° shoulder abduction. Then place finger tips under Pectoralis minor tendon and position the arm in 90°/90° shoulder abduction and elbow flexion. Apply the pressure while stroking the tender area and ask the patient to adduct the arm then bring shoulder backward while maintain the pressure 3 sets of 10 repetition/ 4 days per week for 3 weeks.
  Arms: Experimental interventional group
Other: active control group — Conventional treatment- includes gentle shoulder ROMs i.e. flexion, extension, abduction, adduction, internal rotation and external rotation with-in pain free range, 10 repetitions each for 3 times a day
  Arms: active control group

SUMMARY:
The aim of this research is to determine the Effects of Active Release Technique (ART) on pectoralis minor tightness in post mastectomy women. Randomized controlled trials will be done at Nuclear Medicine, Oncology and Radiotherapy Institute (NORI) Hospital. The sample size will be 60. The subjects were divided in two groups, with 30 subjects in Group A and 30 in Group B. Study duration was of 6 months. Sampling technique applied was Non probability Convenience Sampling technique. Only women aged 40-60 years with Mastectomy (Unilateral/ Bilateral/ Partial/ Radical) and Postoperative chemotherapy/ radiation therapy were included. Tools used in the study are Numeric Pain Rating Score (NPRS), Shoulder Pain and Disability Index (SPADI), Vernier Caliper and Rigid standard plastic transparent right angle. Data was analyzed through SPSS 21.

DETAILED DESCRIPTION:
Breast cancer may be a malignant neoplasm, an abnormal growth (carcinoma) originated in breast tissue that invade the encompassing tissue, grows infiltrative and destructive, and may metastasize.It is outlined pathologically by location of origin within the breast (e.g. ducts, lobes), size of the tumor, standing of the nodes, and also the presence of markers indicating tumor staging. Mostly, early-stage breast cancer diagnosed in women undergo surgical procedures, nearly half withstand breast-conserving surgery and one third experience mastectomy.

It is generally believed that physiotherapy aims to aid recovery and prevent complications following mastectomy however no well-designed, randomized controlled trial has investigated the effect of active release technique (ART) specifically on pectoralis minor in post-operative breast cancer women. Hence, a physiotherapy rehabilitation plan of care consisting of patient education, early mobilization along Active Release Technique (ART) may prevent postoperative complications like chest tightness and reduced shoulder mobility. This will enhance muscular relaxation, improve restricted mobility, and will result in improved quality of life as compared to standard care or conventional treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* women complaining chest tightness
* Mastectomy (Unilateral/ Bilateral/ Partial/ Radical)
* Postoperative chemotherapy or radiation therapy

Exclusion Criteria:

* Tumor Metastasis with other tissue/ organ.
* Underlying Cardiac issues.
* Shoulder joint pathology before surgery.
* Post mastectomy pain syndrome (Pain beyond 3 months).

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only female mastectomy patient will be included
Enrollment: 60 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
NPRS | 3rd week
  Shoulder/Arm pain will assessed using a numerical pain rating scale (NPRS), and scoring range 0, no pain, to 10, maximum pain. pain will be measure from baseline to 1st week to 2nd and 3rd week
Shoulder Pain and Disability Index (SPADI) | 3rd week
  The SPADI is a valid and reliable 13-item shoulder specific instrument measuring both shoulder disability and pain which is divided into two subscales: pain (5 items) and disability (8 items). Scores on both subscales are rated from 0 (no pain or disability) to 10 (worst pain imaginable or so difficult to perform tasks that help is required). The SPADI has proven to be a reliable, valid, and sensitive instrument. Total SPADI score, (0-130), in which, (0-29= little or no pain/disability), (30-49= Mild to moderate pain/disability), (50-130= Moderate to severe pain/disability) It will be measure from baseline to 1st week to 2nd and 3rd week
pectoralis minor length through vernier caliper | 3rd week
  it will be measure from baseline to 1st week to 2nd and 3rd week. Vernier® caliper (intraclass correlation coefficient 0.83-0.87) is used to measure pectoralis minor length. The patients were in the supine position with a normal, relaxed posture. The caliper arms were placed between the coracoid processes to the fourth rib 1-finger apart from lateral to the sternum. As 2.6 cm or 1inch distance has been proposed as the normal length of pectoralis minor muscle
pectoralis minor length through Rigid standard plastic transparent right angle | 3rd week
  it will be measure from baseline to 1st week to 2nd and 3rd week. This tool used to measure the linear distance in millimeter from the table to the posterior acromion of the patients in supine position with the arms by the side and elbows in flexed and rested on abdomen. Without adding any pressure on the table, the base of the protractor was placed on the bed and the vertical side was placed posterior to the acromion

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Federal Breast Cancer Screening center (PIMS), Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No